CLINICAL TRIAL: NCT06367608
Title: Phase 1 Clinical Trial for MR Guided Focused Ultrasound (FUS) Pallidotomy for the Treatment of Task Specific Focal Hand Dystonia (TSFD)
Brief Title: MRgFUS Pallidotomy for the Treatment of Task Specific Focal Hand Dystonia (TSFD)
Acronym: FUS Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Focused Ultrasound Foundation (Other); InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HP-00104695
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Task-Specific Focal Dystonia
MeSH Terms: conditions — Dystonia, Focal, Task-Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ExAblate Transcranial treatment (Experimental): The ExAblate Transcranial system will be used to destroy a small cluster of cells that may be causing the study participant's pain . The ExAblate uses ultrasound to heat a small spot in the brain called globus pallidus internus(GPi). Ultrasound passes through the skin and skull and into the brain to focus on this particular spot.
  Interventions: Device: ExAblate Transcranial treatment

INTERVENTIONS:
Device: ExAblate Transcranial treatment — The ExAblate Transcranial system will be used to destroy a small cluster of cells that may be causing the study participant's dystonia . The ExAblate uses ultrasound to heat a small spot in the brain called globus pallidus internus(GPi). Ultrasound passes through the skin and skull and into the brain to focus on this particular spot.
  Other Names: The ExAblate® MR guided focused ultrasound system

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of MRI-guided focused ultrasound (MRgFUS) for treating task specific focal hand dystonias (TSFD). TSFD is a type of dystonia that affects hand movements during specific tasks such as writing, playing instruments or typing, often causing involuntarily movements or cramping.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and effectiveness of MRI-guided focused ultrasound (MRgFUS) for treating task specific focal hand dystonias (TSFD). TSFD refers to a condition where certain movements or tasks trigger involuntary muscle contractions, particularly during specialized and repetitive activities like writing (known as writer's dystonia), typing (typist's dystonia), playing musical instruments (musician's dystonia), or engaging in sports like golf, table tennis, or juggling. While TSFD affects around 1.2-1.5% of the general population, it's more common among athletes and musicians. Writer's dystonia, for example, typically starts with difficulty writing and hand cramping in the dominant hand, possibly spreading to the arm and shoulder muscles over time. In severe cases, the other hand may also be affected. Similarly, typist's dystonia can lead to finger flexion or extension issues during typing. Musician's dystonia is another form, seen in guitarists, pianists, harpists, or flute players, often emerging during the peak of their careers and significantly impacting musical performance. These dystonias can be career-ending as they impair performance and rarely go into remission, with onset often occurring around the age of forty.

Surgical treatments for Task-Specific Focal Dystonia (TSFD) are less often explored than for other dystonias. Thalamotomy, targeting the ventro-oralis (Vo) nucleus, has shown some promise for hand dystonias like writer's cramp or musician's dystonia. Anecdotally, some benefit from deep brain stimulation (DBS) targeting the globus pallidus internus (GPi) has also been shown, but large-scale studies for TSFD are lacking.

Another promising approach is MR guided focused ultrasound thalamotomy, a non-invasive procedure that uses real-time imaging to precisely target brain areas. This method has already shown success in treating essential tremors and Parkinson's disease symptoms. Recent studies and anecdotal cases have also demonstrated its potential for treating TSFD, with improvements in symptoms observed in patients with writer's cramp, musician's dystonia, and other related conditions.

The Exablate MR Guided Focused Ultrasound Transcranial system is a device designed to overcome the limitations of delivering ultrasound through the intact skull. It uses advanced technology like water-cooling, acoustic correction algorithms, and patient-specific CT data to ensure precise and safe delivery of ultrasound energy to targeted brain areas. This pilot study protocol aims to utilize MR guided focused ultrasound thalamotomy as a treatment option for TSFD.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of moderate to severe TSFD with impact in their daily function or occupation function
2. Patients who failed to response or had unsatisfactory response to the first treatment, such as Botulinum toxin treatment or DBS or refuse these alternative options
3. Age greater than 21 and less than 75 years
4. Subjects who are able and willing to give consent and able to attend all study visits,
5. Documented chronic, symptoms for more than 6 months duration
6. Pallidotomy is feasible based on evaluation of imaging studies
7. Patient able to communicate sensations during the ExAblate TcMRgFUS treatment
8. Two members of the medical team have agreed upon inclusion and exclusion criteria

Exclusion Criteria:

1. Patient with contraindications to MRI such as severe claustrophobia and metallic implants incompatible with MRI.
2. Presence of generalized dystonia or involvement of two or more contiguous body regions (such as Arm along with neck)
3. Severe psychiatric disorder such as uncontrolled depression, anxiety, bipolar disorder, prior attempt at suicide or suicide ideation in preceding 12 months
4. Life expectancy less than 12 months
5. Anticoagulant or antiplatelet medications as well as underlying coagulopathy
6. Pregnant ladies or women of childbearing age who are sexually active and not using contraception
7. Inability to provide informed consent, for example due to underlying cognitive impairment or aphasia
8. Presence of intracranial mass or an acute intracranial abnormality
9. Subjects with unstable cardiac status such as unstable angina pectoris, documented myocardial infarction within 6 months of protocol entry or ejection fraction less than 40
10. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders(DSM-IV)
11. Severe hypertension (diastolic blood pressure > 100 on medication or persistently elevated systolic blood pressure>140 mmHg despite adequate antihypertensive medications)
12. History of intracranial hemorrhage, traumatic brain injury or thalamic stroke.
13. Cerebrovascular disease (multiple cerebrovascular accident's (CVA) or CVA within 6 months)
14. Subjects with life-threatening systemic disease that include and not limited to the following will be excluded from the study participation: HIV, Liver Failure, blood dyscrasias, etc.
15. Subjects with a history of seizures within the past year
16. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hours of total table time.)

    -

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment related adverse events | All events will be reported up to 6 months from treatment
  Procedure related or device related adverse events will be reported, from the treatment day through the 6-month follow-up period.

SECONDARY OUTCOMES:
Change in dystonia intensity | 6 Months
  Efficacy of ExAblate TcMRgFUS for pallidotomy will be evaluated using Arm disability dystonia scale (ADDS) and scales specific to writer's cramp (WCRS) or musician's dystonia (TMDS) scores.
Change in patient's perception of quality of life | 6 months
  Quality of life assessments will be performed with short form (SF)-36 survey
Change in patient's perception of the effect of the procedure | 6 Months
  Patient Global impression of change (PGIC): The effect of the procedure on patient perceived impact of pain related symptoms, emotions and quality of life will be measured using PGIC scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No